CLINICAL TRIAL: NCT04198870
Title: Percutaneous MitraClip Device or Surgical Mitral Valve REpair in PAtients With PrImaRy MItral Regurgitation Who Are Candidates for Surgery (REPAIR MR)
Brief Title: MitraClip REPAIR MR Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-CIP-10304
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Mitral Valve Regurgitation
Keywords: MitraClip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Other): Mitral Valve Repair Surgery
  Interventions: Procedure: Mitral Valve Repair Surgery
- Device Arm (Experimental): MitraClip™ device implantation
  Interventions: Device: MitraClip™ device implantation

INTERVENTIONS:
Device: MitraClip™ device implantation — Transcatheter repair of the mitral valve using MitraClip™ device
  Arms: Device Arm
Procedure: Mitral Valve Repair Surgery — Surgical repair of the mitral valve
  Arms: Control Arm

SUMMARY:
The objective of this randomized controlled trial (RCT) is to compare the clinical outcome of MitraClip™ device versus surgical repair in patients with severe primary MR who are at moderate surgical risk and whose mitral valve has been determined to be suitable for correction by MV repair surgery by the cardiac surgeon on the local site heart team.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has severe (Grade III or greater per the ASE criteria, which includes severity grades of 3+ and 4+) primary MR (mixed etiology is acceptable provided the principal mechanism of action is a degenerative mitral valve) as assessed by the ECL.
2. The cardiac surgeon of the Site Heart Team (consisting of at least one interventionalist, and one cardiac surgeon) has confirmed that the subject is a candidate for mitral valve surgery and the EC have confirmed that the subject's mitral valve anatomy is suitable for percutaneous repair with the MitraClip™ device with high certainty of achieving MR ≤ mild
3. Subject is symptomatic (NYHA Class II/III/IV) or asymptomatic with LVEF ≤ 60%, pulmonary artery systolic pressure > 50 mmHg, or LVESD > 40 mm
4. Subject is at moderate surgical risk defined as being at least 75 years of age at the time of EC review. If younger than 75 years, then the subject should have:

   1. Society of Thoracic Surgeons (STS) Predicted Risk of Mortality (PROM) Repair Score ≥ 2%, OR
   2. Presence of other comorbidities which may introduce a potential surgery-specific impediment
5. Subject provides written informed consent
6. Subject is ≥ 18 years of age

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation
2. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
3. Subject has ischemic or non-ischemic secondary MR
4. Concomitant severe tricuspid valve regurgitation
5. Ejection fraction <30%
6. Severe mitral annular calcification
7. Acute myocardial infarction in the past 12 weeks
8. Need for cardiac surgery to correct pulmonary valve disease, aortic valve disease, or tricuspid valve disease
9. Subjects who have concurrent coronary artery disease that needs to be treated may be included provided the subjects are eligible for both percutaneous coronary intervention (PCI) and coronary artery bypass surgery. Subjects randomized to the device group, must undergo PCI before the MitraClip™ device procedure. Subjects randomized to the surgical (control) arm may undergo coronary artery revascularization during mitral valve repair surgery
10. Surgical procedure performed in the past 30 days
11. Femoral vein cannot accommodate a 24 F catheter or presence of IVC filter would interfere with the catheter or ipsilateral DVT
12. Transesophageal echocardiography (TEE) is contraindicated.
13. Hemodynamic instability: systolic pressure ≤ 90 mmHg without afterload reduction, cardiogenic shock, or the need for inotropic support or IABP
14. Need for emergency surgery for any reason
15. Prior mitral valve surgery, valvuloplasty, mechanical prosthetic valve or VAD
16. Systolic anterior motion of the mitral valve
17. Hypertrophic cardiomyopathy
18. Renal insufficiency requiring dialysis
19. Active infections requiring current antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, stroke, cardiac hospitalization, or acute kidney injury requiring renal replacement therapy at 2 years (any cardiac hospitalizations in the first 30 days post treatment will be excluded) | 2 Years
  The proportion of subjects who are alive, without stroke, CV hospitalization or acute kidney injury requiring renal replacement therapy at 2 years in the Device and Control groups, respectively
Proportion of subjects with moderate or less MR (≤2+), without mitral valve replacement, and without recurrent mitral valve intervention (surgical or percutaneous) | 2 Years
  Proportion of subjects with moderate or less MR (≤2+), without mitral valve replacement, and without recurrent mitral valve intervention (surgical or percutaneous) from the time of index procedure through 2 years in the Device and Control groups, respectively

SECONDARY OUTCOMES:
Proportion of subjects with MR ≤ mild at 30 days post index procedure among survivors | 30 Days
  The proportion of subjects with MR ≤ mild at 30 days post index procedure among survivors will be compared between the Device and Control groups
Number of days at hospital from index procedure to home discharge | At Discharge (≤ 14 days following index procedure)
  Hospital length of stay from index procedure to home discharge (days) in Device group compared to the Control group
Proportion of subjects discharged to home post index hospitalization | At Discharge (≤ 14 days following index procedure)
  The proportion of subjects who are discharged to home post index hospitalization will be compared between the Device and Control groups
Quality of life improvement assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ) of at least 10 points at 2 years compared to baseline among survivors. | 2 Years
  The proportion of subjects who have at least a 10 point improvement in KCCQ at 2 years post index procedure from baseline among survivors will be compared between the Device and Control groups for non-inferiority.
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered questionnaire used for quantifying patient's health status including the symptoms (frequency and burden), physical and social limitations, and quality of life impact due to the heart failure syndrome. Validity, reproducibility, responsiveness and interpretability of the scores have been independently established for each of these health status domains, and overall summary scores are reported in a range of 0-100, in which higher scores reflect better health status.
Severe symptomatic mitral stenosis at 1 year | 1 Year
  The proportion of subjects who have severe symptomatic mitral stenosis at 1 year post index procedure will be compared between the Device and Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCarthy, MD, Principal Investigator — Northwestern Memorial Hospital; Saibal Kar, MD, Principal Investigator — Los Robles Regional Medical Center
Locations (74):
- United States (63):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - St. Josephs Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Scripps Health, La Jolla, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - University of California - Davis Medical Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Saint Joseph Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Medical Center, Jacksonville, Florida
  - NCH Healthcare System, Naples, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Albany Medical Center, Albany, New York
  - South Shore University Hospital, Bay Shore, New York
  - NYU Langone Health, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Rochester Regional Health, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mt. Carmel East, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Pinnacle Health Cardiovascular Institute, Inc., Harrisburg, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Ascension Texas Cardiovascular Research, Austin, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - UTHealth Memorial Hermann, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - The Heart Institute at Virginia Mason, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (4):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Germany (6):
  - Universitätsklinikum Ulm, Ulm, Bad-wur
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Universitätsklinikum Rostock (AöR), Rostock
- Center Inselspital Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] McCarthy PM, Whisenant B, Asgar AW, Ailawadi G, Hermiller J, Williams M, Morse A, Rinaldi M, Grayburn P, Thomas JD, Martin R, Asch FM, Shu Y, Sundareswaran K, Moat N, Kar S. Percutaneous MitraClip Device or Surgical Mitral Valve Repair in Patients With Primary Mitral Regurgitation Who Are Candidates for Surgery: Design and Rationale of the REPAIR MR Trial. J Am Heart Assoc. 2023 Feb 21;12(4):e027504. doi: 10.1161/JAHA.122.027504. Epub 2023 Feb 8. PMID 36752231
- [Derived] Kaneko T, Hirji S, Zaid S, Lange R, Kempfert J, Conradi L, Hagl C, Borger MA, Taramasso M, Nguyen TC, Ailawadi G, Shah AS, Smith RL, Anselmi A, Romano MA, Ben Ali W, Ramlawi B, Grubb KJ, Robinson NB, Pirelli L, Chu MWA, Andreas M, Obadia JF, Gennari M, Garatti A, Tchetche D, Nazif TM, Bapat VN, Modine T, Denti P, Tang GHL; CUTTING-EDGE Investigators. Mitral Valve Surgery After Transcatheter Edge-to-Edge Repair: Mid-Term Outcomes From the CUTTING-EDGE International Registry. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2010-2021. doi: 10.1016/j.jcin.2021.07.029. PMID 34556275